CLINICAL TRIAL: NCT00587678
Title: Comprehensive Magnetic Resonance of Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christopher M. Kramer MD, Professor of Radiology and Medicine, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10387; R01HL075792 (NIH)
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2012-02-03 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Peripheral Artery Disease
Keywords: PAD
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Simvastatin; Ezetimibe; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Randomized (Experimental): Patients are imaged at baseline and randomized to Simvistatin 40 mg each night or Simvistatin 40mg/Zetia 10mg each night for 2 years
  Interventions: Drug: Simvastatin; Drug: Simvastatin/Ezetimibe
- Ezetemibe (Experimental): Patients are imaged at baseline and treated with ezetimibe 10mg each night for 2 years.
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Simvastatin — 40mg each night
  Other Names: Zocor
  Arms: Randomized
Drug: Ezetimibe — 10mg daily
  Other Names: Zetia
  Arms: Ezetemibe
Drug: Simvastatin/Ezetimibe — 40mg/10mg each night
  Other Names: Vytorin
  Arms: Randomized

SUMMARY:
The purpose of this study is to develop new ways of imaging fatty blockages in the leg arteries to improve upon techniques used now and to develop new ways of understanding how new treatments may affect the disease.

ELIGIBILITY:
Inclusion Criteria:

Patients age 30-85 referred to the vascular imaging laboratory with documented evidence of peripheral arterial disease (0.4<ABI<0.9) 96 Normal healthy subjects ages 30-85

Exclusion Criteria:

Age<30, >85

GFR less than 45mL/min based on a serum creatinine drawn within 90 days of the MRI:

Pregnancy Contraindications to a magnetic resonance examination

* Intracranial clips
* Implantable pacemaker and defibrillator
* Cochlear or intraocular implants
* Claustrophobia
* Any metallic implant not listed as magnetic resonance compatible in Shellock F.G ---Pocket Guide to Magnetic Resonance Procedures and Metallic Objects, Update 2000. Lippincott, Williams and Wilkins

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2006-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Kramer, M.D., Principal Investigator — University of Virginia Health System
Locations (1):
- University of Virgina Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Isbell DC, Berr SS, Toledano AY, Epstein FH, Meyer CH, Rogers WJ, Harthun NL, Hagspiel KD, Weltman A, Kramer CM. Delayed calf muscle phosphocreatine recovery after exercise identifies peripheral arterial disease. J Am Coll Cardiol. 2006 Jun 6;47(11):2289-95. doi: 10.1016/j.jacc.2005.12.069. Epub 2006 May 15. PMID 16750698
- [Background] Isbell DC, Meyer CH, Rogers WJ, Epstein FH, DiMaria JM, Harthun NL, Wang H, Kramer CM. Reproducibility and reliability of atherosclerotic plaque volume measurements in peripheral arterial disease with cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2007;9(1):71-6. doi: 10.1080/10976640600843330. PMID 17178683
- [Background] Isbell DC, Epstein FH, Zhong X, DiMaria JM, Berr SS, Meyer CH, Rogers WJ, Harthun NL, Hagspiel KD, Weltman A, Kramer CM. Calf muscle perfusion at peak exercise in peripheral arterial disease: measurement by first-pass contrast-enhanced magnetic resonance imaging. J Magn Reson Imaging. 2007 May;25(5):1013-20. doi: 10.1002/jmri.20899. PMID 17410566
- [Background] Kramer CM. Peripheral arterial disease assessment: wall, perfusion, and spectroscopy. Top Magn Reson Imaging. 2007 Oct;18(5):357-69. doi: 10.1097/rmr.0b013e31815d064c. PMID 18025990
- [Result] West AM, Anderson JD, Meyer CH, Epstein FH, Wang H, Hagspiel KD, Berr SS, Harthun NL, DiMaria JM, Hunter JR, Christopher JM, Chew JD, Winberry GB, Kramer CM. The effect of ezetimibe on peripheral arterial atherosclerosis depends upon statin use at baseline. Atherosclerosis. 2011 Sep;218(1):156-62. doi: 10.1016/j.atherosclerosis.2011.04.005. Epub 2011 Apr 16. PMID 21570685
- [Result] West AM, Anderson JD, Epstein FH, Meyer CH, Wang H, Hagspiel KD, Berr SS, Harthun NL, Weltman AL, Dimaria JM, Hunter JR, Christopher JM, Kramer CM. Low-density lipoprotein lowering does not improve calf muscle perfusion, energetics, or exercise performance in peripheral arterial disease. J Am Coll Cardiol. 2011 Aug 30;58(10):1068-76. doi: 10.1016/j.jacc.2011.04.034. PMID 21867844
- [Derived] Anderson JD, Epstein FH, Meyer CH, Hagspiel KD, Wang H, Berr SS, Harthun NL, Weltman A, Dimaria JM, West AM, Kramer CM. Multifactorial determinants of functional capacity in peripheral arterial disease: uncoupling of calf muscle perfusion and metabolism. J Am Coll Cardiol. 2009 Aug 11;54(7):628-35. doi: 10.1016/j.jacc.2009.01.080. PMID 19660694

RESULTS

PARTICIPANT FLOW:
Groups:
- Simvastatin 40mg: Statin naive patients randomized to simvastatin 40mg qhs after baseline studies for 2 years
- Simvastatin 40mg/Ezetimibe 10 mg: Statin naive patients randomized to simvastatin 40mg/Ezetimibe 10mg qhs after baseline studies for 2 years
- Ezetimibe 10mg: Open label Ezetimibe 10mg daily begun after baseline studies for 2 years
Period: Overall Study
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg
Started | 22 | 22 | 41
Completed | 16 | 18 | 33
Not Completed | 6 | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg | Total
Number analyzed (Participants) | 22 | 22 | 41 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 11 | 20 | 47
  >=65 years | 6 | 11 | 21 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12) | 64 (9) | 66 (11) | 63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 21 | 37
  Male | 16 | 12 | 20 | 48
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 41 | 85
Total cholesterol [Mean (Standard Deviation); unit: mg/dl] | 194 (11) | 189 (10) | 170 (6) | 182 (45)
Low density lipoprotein cholesterol [Mean (Standard Deviation); unit: mg/dl] | 118 (10) | 118 (9) | 100 (4) | 111 (35)
High density lipoprotein cholesterol [Mean (Standard Deviation); unit: mg/dl] | 45 (4) | 48 (4) | 42 (2) | 43 (13)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 227 (47) | 130 (21) | 157 (20) | 159 (104)
Plaque volume [Mean (Standard Deviation); unit: cm^3] | 11.0 (1.5) | 11.5 (1.4) | 10.0 (0.8) | 10.6 (5.4)
Total vessel volume [Mean (Standard Deviation); unit: cm^3] | 17.7 (2.5) | 17.5 (2.4) | 15.7 (1.2) | 16.6 (8.7)
Lumen volume [Mean (Standard Deviation); unit: cm3] | 6.7 (1.2) | 5.9 (1.1) | 5.7 (0.5) | 6.0 (3.8)
Perfusion index [Mean (Standard Deviation); unit: Units on a scale (0 = worst, 1 = best).] — First pass contrast-enhanced MRI measure of exercise calf muscle perfusion
  Units on a scale (0 = worst, 1 = best). | 0.48 (0.18) | 0.42 (0.13) | 0.51 (0.16) | 0.48 (0.16)
Phosphocreatine recovery time constant [Mean (Standard Deviation); unit: seconds] — Phosphocreatine recovery time constant measured at peak exercise with 31P magnetic resonance spectroscopy. The range is from 20 to 1000 seconds with 20-40 being normal and higher than 40 abnormal.
  seconds | 94 (77) | 104 (56) | 83 (62) | 92 (64)
Magnetic resonance angiographic index [Mean (Standard Deviation); unit: units on a scale (0-4). 0 = normal.] — Index of stenoses based on MR angiogram (0=normal, 4=worst possible)
  units on a scale (0-4). 0 = normal. | 0.73 (0.50) | 1.10 (0.72) | 0.65 (0.62) | 0.81 (0.64)
Log of Treadmill Exercise Time [Mean (Standard Deviation); unit: log of time in seconds] | 6.08 (0.84) | 5.82 (0.67) | 5.94 (0.78) | 5.95 (0.76)
6-minute walk distance [Mean (Standard Deviation); unit: feet] | 1103 (407) | 976 (324) | 1007 (435) | 1024 (397)
V02 max - maximal oxygen consumption [Mean (Standard Deviation); unit: ml/kg/min] — Measured during treadmill exercise
  ml/kg/min | 14.6 (4.6) | 12.4 (3.2) | 12.1 (3.8) | 12.8 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Plaque Volume
Description: SFA plaque volume
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg
Number analyzed (Participants) | 16 | 18 | 33
cm^3 | 10.5 (1.4) | 10.5 (1.3) | 10.8 (0.9)
Statistical Analysis 1: Comparison: Simvastatin 40mg vs Simvastatin 40mg/Ezetimibe 10 mg; Test type: Superiority or Other; p = 0.32, Linear repeated measures model
Statistical Analysis 2: Comparison: Ezetimibe 10mg; Test type: Superiority or Other; p < 0.01, Linear repeated measures model — vs. baseline

2. Secondary Outcome: Low Density Lipoprotein Cholesterol
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg
Number analyzed (Participants) | 16 | 18 | 33
mg/dl | 83 (11) | 68 (10) | 77 (5)
Statistical Analysis 1: Comparison: Simvastatin 40mg vs Simvastatin 40mg/Ezetimibe 10 mg; Test type: Superiority or Other; p = 0.31, Linear repeated measures model
Statistical Analysis 2: Comparison: Ezetimibe 10mg; Test type: Superiority or Other; p < 0.05, Linear repeated measures model — vs. baseline

3. Primary Outcome: Perfusion Index
Description: Perfusion index is a MRI measure of calf muscle perfusion indexed to the arterial input. The value is between 0 and 1 with 0 being worst and 1 being best.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Units on a scale (0 = worst, 1 = best)
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg
Number analyzed (Participants) | 16 | 18 | 33
Units on a scale (0 = worst, 1 = best) | 0.34 (0.19) | 0.37 (0.13) | 0.54 (0.20)
Statistical Analysis 1: Comparison: Simvastatin 40mg vs Simvastatin 40mg/Ezetimibe 10 mg vs Ezetimibe 10mg; Test type: Superiority or Other; p = 0.71, Linear repeated measures model

4. Primary Outcome: Phosphocreatine Recovery Time Constant - the Time it Takes for Phosphocreatine Levels to Recover to Plateau.
Description: Phosphocreatine recovery time constant is the time it takes for phosphocreatine levels to recover to plateau after the completion of exercise. This ranges from 20 to 1000 seconds. 20-40 seconds is normal and any value over 40 seconds is abnormal.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg
Number analyzed (Participants) | 16 | 18 | 33
seconds | 84 (68) | 73 (35) | 74 (58)
Statistical Analysis 1: Comparison: Simvastatin 40mg vs Simvastatin 40mg/Ezetimibe 10 mg vs Ezetimibe 10mg; Test type: Superiority or Other; p = 0.67, Linear repeated measures model

5. Secondary Outcome: Total Cholesterol
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg
Number analyzed (Participants) | 16 | 18 | 33
mg/dl | 152 (12) | 136 (12) | 144 (6)
Statistical Analysis 1: Comparison: Simvastatin 40mg vs Simvastatin 40mg/Ezetimibe 10 mg; Test type: Superiority or Other; p = 0.37, Linear repeated measures model
Statistical Analysis 2: Comparison: Ezetimibe 10mg; Test type: Superiority or Other; p < 0.05, Linear repeated measures model — vs. baseline

6. Secondary Outcome: High Density Lipoprotein Cholesterol
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg
Number analyzed (Participants) | 16 | 18 | 33
mg/dl | 44 (4) | 46 (3) | 43 (3)
Statistical Analysis 1: Comparison: Simvastatin 40mg vs Simvastatin 40mg/Ezetimibe 10 mg vs Ezetimibe 10mg; Test type: Superiority or Other; p = 0.78, Linear repeated measures model

7. Secondary Outcome: Triglycerides
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg
Number analyzed (Participants) | 16 | 18 | 33
mg/dl | 171 (30) | 119 (20) | 152 (15)
Statistical Analysis 1: Comparison: Simvastatin 40mg vs Simvastatin 40mg/Ezetimibe 10 mg vs Ezetimibe 10mg; Test type: Superiority or Other; p = 0.68, Linear repeated measures model

8. Secondary Outcome: Magnetic Resonance Angiographic Index
Description: MRA index is a measure of angiographic severity of disease. 0 = no disease and 4 is severe disease.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: units on scale (0 = normal, 4 = worst)
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg
Number analyzed (Participants) | 16 | 18 | 33
units on scale (0 = normal, 4 = worst) | 0.71 (0.46) | 1.32 (0.86) | 0.63 (0.64)
Statistical Analysis 1: Comparison: Simvastatin 40mg vs Simvastatin 40mg/Ezetimibe 10 mg; Test type: Superiority or Other; p < 0.05, Linear repeated measures model

9. Secondary Outcome: Log Treadmill Exercise Time
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: log time in seconds
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg
Number analyzed (Participants) | 16 | 18 | 33
log time in seconds | 5.92 (1.08) | 5.79 (0.67) | 5.78 (0.63)
Statistical Analysis 1: Comparison: Simvastatin 40mg vs Simvastatin 40mg/Ezetimibe 10 mg vs Ezetimibe 10mg; Test type: Superiority or Other; p = 0.67, linear repeated measures model

10. Secondary Outcome: 6-minute Walk Distance
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: ft.
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg
Number analyzed (Participants) | 16 | 18 | 33
ft. | 1078 (485) | 1038 (248) | 1099 (394)
Statistical Analysis 1: Comparison: Simvastatin 40mg vs Simvastatin 40mg/Ezetimibe 10 mg vs Ezetimibe 10mg; Test type: Superiority or Other; p = 0.77, Linear repeated measures model

11. Secondary Outcome: V02 - Maximal Oxygen Consumption
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: ml/min/kg
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg
Number analyzed (Participants) | 16 | 18 | 33
ml/min/kg | 14.8 (4.6) | 12.1 (2.9) | 12.3 (4.6)
Statistical Analysis 1: Comparison: Simvastatin 40mg vs Simvastatin 40mg/Ezetimibe 10 mg vs Ezetimibe 10mg; Test type: Superiority or Other; p = 0.85, Linear repeated measures model

ADVERSE EVENTS:
Arm/Group | Simvastatin 40mg | Simvastatin 40mg/Ezetimibe 10 mg | Ezetimibe 10mg
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22 | 0/41
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No